CLINICAL TRIAL: NCT05620771
Title: Phase II Study Therasphere® (Yttrium-90) in Combination With Systemic Therapy in Patients With High-risk Hepatocellular Carcinoma
Brief Title: Therasphere® and Systemic Therapy for Patients With Hepatocellular Carcinoma That is High-risk
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Per PI request
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 22I07; NCI-2022-09476 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA060553 (NIH); NU 22I07 (Other: Northwestern University)
Record Dates: First submitted 2022-11-11; First posted 2022-11-17 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab; Yttrium-90

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Y90 + Atezolizumab and Bevacizumab (Experimental)
  Interventions: Drug: Atezolizumab and Bevacizumab
- Y90 + TKI (Experimental)
  Interventions: Drug: Y90 + TKI

INTERVENTIONS:
Drug: Atezolizumab and Bevacizumab — Patients will receive atezolizumab + Bevacizumab for 21 days after standard of care therapy is complete.
  Arms: Y90 + Atezolizumab and Bevacizumab
Drug: Y90 + TKI — Patients will receive TKI for 21 days after standard of care therapy is complete.
  Arms: Y90 + TKI

SUMMARY:
The purpose of this research is to compare progression free survival between two available systemic therapies - immunotherapy and tyrosine kinase inhibitors - after Therasphere® (yttrium-90) treatment in adult patients with advanced hepatocellular carcinoma. The immunotherapy consists of a standard-of-care treatment with Atezolizumab and Bevacizumab. Treatment with tyrosine kinase inhibitors consists of standard-of-care Lenvatinib or Cabozantinib.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare Progression Free Survival (PFS) in patients with advanced HCC who receive Y90 followed by immunotherapy (atezolizumab + bevacizumab, Arm A) or Y90 followed by TKI treatment ( lenvatinib or cabozantinib, Arm B). For ARM B, [patients will receive Lenvatinib. If they have prior history of treatment with Lenvatinib, then can be given Cabozantinib]..

SECONDARY OBJECTIVES:

I. To compare the Time to Progression (TTP) in patients with advanced HCC who receive Immunotherapy combination compared to TKI following Y90.

II. To compare the Objective Response Rate (ORR) as assessed by RECIST v1.1 in patients with advanced HCC who receive immunotherapy combination and those who receive TKI treatment after Y90.

III. To compare the Duration of Response (DOR) in patients with advanced HCC who receive immunotherapy combination and those who receive TKI treatment after Y90.

IV. To compare the Clinical Benefit Rates (CBR) [CR, PR,SD] as assessed by RECIST v1.1 in patients with advanced HCC who receive immunotherapy combination and those who receive TKI treatment after Y90.

V. To compare the Overall Survival (OS) in patients with advanced HCC who receive immunotherapy combination and those who receive TKI treatment after Y90.

VI. To compare the safety and tolerability of patients with advanced HCC who receive immunotherapy combination and those who receive TKI treatment after Y90, as defined by NCI CTCAEv5.

OUTLINE:

Patients will first be treated one time with liver directed therapy, Therasphere® (Y-90), following institutional procedures. After completion of Y- 90, patients will have some recovery time (14-21 days) prior to starting systemic therapy.

Patients will be followed up for 2 years after completion of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of hepatocellular carcinoma (HCC) confirmed by American Association for Study of Liver Diseases (AASLD) guidelines with a Childs-Pugh score of A or B7 NOTE: If the patient does not have histological confirmation of disease by biopsy, diagnosis of HCC must be documented with approval by a tumor board or other multidisciplinary conference. Please refer to the appropriate source documents.
* Patients must have at least 1 lesion that is measurable using RECIST guidelines. NOTE: A previously irradiated lesion can be considered a target lesion if the lesion is well defined, measurable per RECIST, and has clearly progressed.
* Patients must have advanced disease that is not amenable to transplant or resection.
* Patients may be treatment naïve or have received any number of prior therapies. NOTE:

Prior cancer targeted immunotherapy is contraindicated and not permitted.

* Patients must exhibit an ECOG performance status of 0, 1, or 2 [Appendix 1]
* Patients must have adequate organ function prior to registration as determined by:
* Adequate organ function parameters:

  1. HEMATOLOGICAL (without growth factor support)

     * Hemoglobin (HgB) ≥ 8.5 g/dL (without the use of growth factors) [transfusion permitted]
     * Absolute Neutrophil Count (ANC) ≥1000 microliter (µL)
     * Platelet Count ≥ 50 x 109/L (without use of growth factors [i.e., IL-11 ] [Transfusion permitted to achieve this value]
     * Prothrombin time (PT)/ International normalized ratio (INR)
     * NOTE: Subjects receiving anticoagulant therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation. ≤ 2.3 or PT ≤ 6 seconds above control.
  2. RENAL

     • Calculated creatinine clearance (*Cockcroft-Gault formula will be used to calculate CrCl)[Appendix 2] (CrCl) or 24-hour urine CrCl > 30 mL/min
  3. HEPATIC

     * Serum Bilirubin ≤ 3 times the upper limit of normal (ULN)
     * AST ≤ 5 times ULN
     * ALT ≤ 5 times ULN Abbreviations: ALT = alanine aminotransferase; ANC = absolute neutrophil count; AST = aspartate aminotransferase; ULN = upper limit of normal.
* For patients with a known history of Human immunodeficiency virus (HIV), infected patients on effective anti-retroviral therapy
* For patients with a known history of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a known history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligibleif they have an undetectable HCV viral..
* Females of childbearing potential (FOCBP), and non-sterilized males who are sexually active must agree to the use of two methods of contraception, with one method being highly effective and the other method being either highly effective or less effective. They must also refrain from egg and/or sperm cell donation and breastfeeding for 90 days after the final dose of investigational product(s) FOCBP are defined as those who are not surgically sterile (i.e. bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause) FOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment. .

Men who are sexually active with FOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment.

* FOCBP must have a negative pregnancy test (Serum or urine pregnancy test per site investigator discretion) within 7 days prior to registration.
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study.

Exclusion Criteria:

* Patients who are concurrently enrolled in another clinical study unless it is an observational (non- interventional) clinical study or the follow-up period of an interventional study.
* Patients who are receiving any other investigational agents within 28 days of registration.
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to Y90, PD-1 &PD-L1 antagonists and TKI's.

Note: Patients must not have a history of severe allergic reactions (i.e., Grade 4 allergy, anaphylactic reaction from which the subject did not recover within 6 hours of institution of supportive care) to any unknown allergens or any components of the systemic therapy

* Patients must not have had prior treatment any PDL1 or PD-1 antagonists
* Patients who have known additional malignancy that progressed or required treatment within the last 3 years. Exceptions include adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for at least three years.
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including chronic prolonged systemic corticosteroids (defined as corticosteroid use of duration one month or greater), should be excluded. These include but are not limited to patients with a history of: immune related neurologic disease

  * multiple sclerosis
  * autoimmune (demyelinating) neuropathy NU22I07 10.25.22 initial 19
  * Guillain-Barre syndrome
  * myasthenia gravis
  * systemic autoimmune disease such as SLE
  * connective tissue diseases
  * scleroderma
  * inflammatory bowel disease (IBD)
  * Crohn's
  * ulcerative colitis
  * patients with a history of toxic epidermal necrolysis (TEN)
  * Stevens-Johnson syndrome
  * anti-phospholipid syndrome NOTE: Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Patients with renal failure currently requiring dialysis of any kind .
* Patients with untreated central nervous system (CNS) metastatic disease (including spinal cord and leptomeningeal disease) are excluded.

Note: Subjects with previously treated CNS metastases that are radiographically and neurologically stable for at least 6 weeks and do not require corticosteroids (of any dose) for symptomatic management are permitted to enroll

* Patients receiving any concurrent chemotherapy, biologic or hormonal therapy for cancer treatment within 28 days of registration. Note: Prior cancer immunotherapy is not permitted. Note: Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable.
* Patients who have unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v 5 [Appendix 6] Grade 0 or 1 with the exception of alopecia and laboratory values listed per the inclusion criteria. Note: Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by any of the investigational products may be included (e.g., hearing loss) after consultation with the PI and NU QAM.
* Patients receiving radiation therapy within 14 days of registration.
* Patients receiving live vaccines within 28 days of study registration.
* No systemic glucocorticoids will be permitted within 48 hours prior to study registration.

Note: Topical steroids, bronchodilators and local steroid injections are permitted if clinically required.

* Patients with cardiac disease defined as one of the following are not eligible:

  * Congestive heart failure > class II NYHA.[Appendix 4]
  * Unstable angina (anginal symptoms at rest) or new onset angina (began within the last 90 days )
  * Myocardial infarction within the past 180 days.
* Patients with cardiac ventricular arrhythmias requiring anti-arrhythmic therapy .
* Patients having elevated lung shunting precluding treatment with Y-90.
* Patients who have had major surgery within 4 weeks prior to registration.
* Patients with a history of gastrointestinal bleeding (GIB) within 6 weeks prior to registration.
* Patients with prior transplant of any kind
* Patients who are pregnant or nursing .
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Hypertension that is not controlled on medication
  * Patients who have active clinically serious infection > CTCAEv 5 Grade 2 . Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
  * Active alcohol use, drug use, or a psychiatric disease that would, in the opinion of the PI or a sub-investigator (sub-I), prevent the subject from complying with the study protocol and/or endanger the subject during their participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 2 years
  To compare PFS by RECIST v1.1 criteria, with Y90 followed by immunotherapy (atezolizumab + bevacizumab, Arm A) or Y90 followed by TKI treatment (lenvatinib or cabozantinib, Arm B). Progression is defined as either radiological progression (with MRI or CT scan) OR clinical progression.

SECONDARY OUTCOMES:
Time to Progression (TTP) | Up to 2 years
  To compare the TTP in patients with advanced HCC who receive Immunotherapy combination compared to TKI following Y90. The TTP will be measured as the time of the last available radiographical or clinical disease assessment documenting lack of disease progression.
Objective Response Rate (ORR) | Up to 2 years
  To compare the ORR as assessed by RECIST v1.1 in patients with advanced HCC who receive immunotherapy combination and those who receive TKI treatment after Y90. This will be assessed based on imaging.
Duration of Response (DOR) | Up to 2 years
  To compare the DOR in patients by RECIST v1.1 criteria and is defined as either radiological progression (with MRI or CT scan) OR clinical progression.
Clinical Benefit Rates (CBR) | Up to 2 years
  To compare the CBR as assessed by RECIST v1.1, CBR is defined as the percentage of patients with best response documented as Complete Response (CR), plus those with Partial Response (PR) plus those with Stable Disease (SD).
Overall Survival (OS) | Up to 2 years
  OS is defined from the date of randomization to the study until the date of death from any cause for up to 2 years.
Adverse Events | Up to 2 years
  To compare the safety and tolerability of patients with advanced HCC who receive immunotherapy combination and those who receive TKI treatment after Y90, as defined by NCI CTCAEv5.

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Kalyan, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States